CLINICAL TRIAL: NCT00386191
Title: Evaluation of the Safety and Efficacy of Clopidogrel sulfate50mg and Clopidogrel Sulfate 75mg for the Treatment of Cerebral Infarction
Brief Title: Safety and Efficacy of Clopidogrel for Cerebral Infarction Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SFY6913; SR25990
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2010-02

CONDITIONS: Cerebral Infarction
Keywords: Platelet Aggregation Inhibitors; Ischemic cerebrovascular disease
MeSH Terms: conditions — Cerebral Infarction | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): 50 mg
  Interventions: Drug: clopidogrel (SR25990C)
- 2 (Experimental): 75 mg
  Interventions: Drug: clopidogrel (SR25990C)

INTERVENTIONS:
Drug: clopidogrel (SR25990C) — oral administration

SUMMARY:
The primary objective is to compare the safety of clopidogrel 50mg and 75mg in cerebral infarction with respect to incidence of bleeding adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an episode of cerebral infarction (excluding cardiogenic cerebral thromboembolism) occurring at least 8 days prior to randomization and for whom the clinical course up to randomization is well-documented
* Patients with a cerebral infarct confirmed by Computed Tomography or Magnetic Resonance Image
* Body weight : > 50 kg

Exclusion Criteria:

* Patients with cardiogenic cerebral thromboembolism or disease that could precipitate cardiogenic cerebral thromboembolism, such as atrial fibrillation or valvular hear disease (including valve replacement)
* Patients with Transient Ischemic Attack occuring after the last episode of cerebral infarction
* Patients with serious impairment that would hinder detection of new ischemic event
* Patients with bleeding diathesis, coagulopathy, or hemorrhagic disease
* Patients with history of intracranial hemorrhage
* Patients with diabetic retinopathy
* Hypertensive patients with a persistent increase of blood pressure.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1110 (Actual)
Dates: Start 2006-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Incidence of bleeding adverse events | study period

SECONDARY OUTCOMES:
Incidence of Serious Adverse Events, serious bleeding events, adverse events. Incidence of vascular events. | study period

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Tokyo, Japan